CLINICAL TRIAL: NCT03548545
Title: Trancranial Direct Current Stiimulation as add-on Treatment to Cognitive-Behavior Therapy in People With Major Depression
Brief Title: tDCS as add-on Treatment to Cognitive-Behavior Therapy in People With MDD
Acronym: ESAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Minho (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Sandra Carvalho, PhD, University of Minho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SECVS 174/2017
Record Dates: First submitted 2018-03-28; First posted 2018-06-07 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Major Depressive Disorder; CBT; Transcranial Direct Current Stimulation
Keywords: MDD; CBT; tDCS
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: This is a parallel randomized, double blinded, sham controlled clinical trial in which a total of 72 MDD subjects(36 per arm) will be randomized to one of two groups: CBT combined with either active or sham tDCS.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Both the Participant, the outcome assessor and the Psychologist providing the CBT will be blinded to the type of the stimulation that the subject is receiving. Unblinding will occur at the end of the participation in the study and subjects that received sham tDCS will have the chance to receive the active tDCS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT combined with active tDCS (Experimental): Subjects allocated to this arm will receive cognitive-behavior therapy combined with active tDCS over the dorsolateral prefrontal cortex.
  Interventions: Device: tDCS
- CBT combined with sham tDCS (Sham Comparator): Subjects allocated to this arm will receive cognitive-behavior therapy combined with sham tDCS over the dorsolateral prefrontal cortex.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — subjects will receive a total of 8-structured CBT sessions administered by a certified therapist(according to the NICE guidelines).In the first two weeks, participants will undergo 6-sessions of CBT every other day(3 CBT sessions per week) and 10 daily sessions of either active or sham tDCS(2 mA, 30 minutes).They will undergo additional booster sessions of the same intervention(active or sham tDCS followed by CBT) by week 4 and 6.
  Other Names: CBT

SUMMARY:
This is a parallel randomized, double-blinded, sham-controlled clinical trial in which a total of 72 drug-naïve MDD subjects (36 per arm) are randomized to one of two groups: Cognitive-Behavior Therapy (CBT) combined with either active or sham tDCS.

The primary outcome is mood improvement, as measured by the Montgomery-Asberg Depression Rating Scale (MADRS). The secondary outcome is to test whether tDCS combined with CBT can engage the proposed mechanistic target, of restoring the prefrontal imbalance and connectivity, by changes over EEG.

DETAILED DESCRIPTION:
Major Depression Disorder (MDD) is widely recognized as a staggering global healthcare challenge, as well as a potentially lethal illness. In Portugal, 7% of the population is diagnosed with depression every year, and suicide is responsible for more than a thousand deaths annually.

The current standard care for MDD involves the use of psychotherapy, antidepressant medication, or a combination of both. However, approximately 30% of people suffering from MDD exhibit depressive symptoms despite the appropriate psychological and pharmacological treatments. One option is to combine several treatments, usually by the use of drug augmentations and/or combinations of different drugs, which often increases the risk of adverse effects. Thus, it is important to study non-pharmacological interventions targeting mechanisms not directly involved with the regulation of neurotransmitters.

Cognitive-behavioral Therapy (CBT) is a well-established, and empirically-supported non-pharmacological treatment for depression, including for those that have not responded to antidepressants. However, several patients remain refractory to CBT.

tDCS is a safe, non-invasive, rather inexpensive, easy to administrate, and well-tolerated neuromodulatory technique. Several studies, including studies from our group, already shown that tDCS can be effective in MDD. However, tDCS seems to have a better effect when used as an add-on treatment to other intervention.

What is not known so far are the effects of using tDCS as add-on intervention to CBT on MDD symptoms.

Therefore, this is a parallel randomized, double-blinded, sham-controlled clinical trial in which a total of 72 first-episode MDD subjects (36 per arm) will be randomized to one of two groups: CBT combined with either active or sham tDCS. The design and the tDCS parameters will be similar to the SELECT trial by Brunoni et al. (2013).

The primary outcome is mood improvement, as measured by the Montgomery-Asberg Depression Rating Scale (MADRS). The secondary outcome is to test whether tDCS combined with CBT can engage the proposed mechanistic target, of restoring the prefrontal imbalance and connectivity, by changes over resting-state EEG and fMRI.

ELIGIBILITY:
Inclusion Criteria:

* 1)Aged 18-75 years;
* 2)Unipolar, nonpsychotic MDD;
* 3)Score in the MADRS between 7 and 34(mild to moderate depression);
* 4)Low risk of suicide;
* 5)Able to sign informed consent

Exclusion Criteria:

* 1)Any contraindication to receive tDCS(such as metal in the head, implanted brain medical devices);
* 2)any significant or unstable neurologic or psychiatric disorder other than MDD;2) history of substance abuse within the past 6-months;
* 3)Any personality disorders; and
* 5)any severe life-threatening Axis III disorders or concurrent medical condition likely to worsen patient's functional status in next 6-months such as; cancer, terminal heart, kidney, or liver disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2018-03-28 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Mood improvement | Improvement defined as 50% decrease in the MADRS score at 4-week intervention. Cut-off points include: 0 to 6 - symptom absent, 7 to 19 - mild depression, 30 to 34 - moderate, 35 to 60 - severe depression.
  Mood as assessed by the Montgomery-Asberg Depression Rating Scale(MADRS)

SECONDARY OUTCOMES:
EEG activity | Reduction of the inter-hemispheric imbalance over DLPFC at 4-week post-intervention sessions
  EEG alpha activity over the prefrontal cortex

CONTACTS AND LOCATIONS:
Overall Officials: Sandra R Carvalho, PhD, Principal Investigator — Cipsi, School of Psychology, University of Minho
Locations (1):
- School of Psychology, University of Minho, Braga, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Carvalho S, Goncalves OF, Brunoni AR, Fernandes-Goncalves A, Fregni F, Leite J. Transcranial Direct Current Stimulation as an Add-on Treatment to Cognitive-Behavior Therapy in First Episode Drug-Naive Major Depression Patients: The ESAP Study Protocol. Front Psychiatry. 2020 Nov 3;11:563058. doi: 10.3389/fpsyt.2020.563058. eCollection 2020. PMID 33240121